CLINICAL TRIAL: NCT00791219
Title: A Randomized, Double Blind, Multiple-site, Placebo-Controlled Study, Comparing the Efficacy and Safety of SUBA™-Itraconazole Capsules Compared to SPORANOX® (Itraconazole) Capsules in the Treatment of Onychomycosis of the Toenail
Brief Title: Study Comparing SUBA™-Itraconazole With SPORANOX® (Itraconazole) in the Treatment of Onychomycosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Halcygen Pharmaceuticals Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 70850702; HGN06 (Other: Halcygen Pharmaceuticals)
Record Dates: First submitted 2008-11-12; First posted 2008-11-14 (Estimated); Results first posted 2020-08-25 (Actual); Last update posted 2020-08-25 (Actual); Status verified 2020-08

CONDITIONS: Onychomycosis
Keywords: Onychomycosis
MeSH Terms: conditions — Onychomycosis | interventions — Itraconazole

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Test (Experimental): 100 mg approximately 30 minutes prior to breakfast for 12 weeks of SUBA™-Itraconazole 50 mg capsules (HalcyGen Ltd)
  Interventions: Drug: SUBA-itraconazole
- Reference (Active Comparator): 200 mg taken with breakfast of SPORANOX® (itraconazole) 100 mg capsules (Janssen Pharma).
  Interventions: Drug: Itraconazole
- Placebo (Placebo Comparator): Two placebo capsules taken approximately 30 minutes prior to breakfast
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SUBA-itraconazole — 100 mg approximately 30 minutes prior to breakfast for 12 weeks of SUBA™-Itraconazole 50 mg capsules (HalcyGen Ltd)
  Other Names: itraconazole 50 mg capsules
  Arms: Test
Drug: Itraconazole — 200 mg taken with breakfast of SPORANOX® (itraconazole) 100 mg capsules (Janssen Pharma).
  Other Names: Sporanox
  Arms: Reference
Drug: Placebo — Two placebo capsules taken approximately 30 minutes prior to breakfast
  Other Names: placebo capsules
  Arms: Placebo

SUMMARY:
The objective of this study is to compare the relative efficacy and safety of SUBA™-Itraconazole Capsules (HalcyGen Ltd) to an already marketed oral formulation of itraconazole SPORANOX® (itraconazole) capsules (Janssen Pharma) in the treatment of onychomycosis of the toenail. Both the test and the reference formulations will also be compared to a placebo formulation to test for superiority.

DETAILED DESCRIPTION:
Randomized, Double-Blind, Multiple-Site, Placebo-Controlled, Parallel designed study comparing a dosing regimen of 100 mg approximately 30 minutes prior to breakfast for 12 weeks of SUBA™-Itraconazole 50 mg capsules (HalcyGen Ltd) to the approved dosing regimen of 200 mg taken with breakfast of SPORANOX® (itraconazole) 100 mg capsules (Janssen Pharma). Patients will be randomly assigned in a 3:3:1 ratio to the test product 100 mg once-a-day: reference product 200 mg once-a-day: placebo once-a-day. respectively. The patients will complete 5 visits: baseline/screening (within 28 days of randomization), Day 1 (randomization), Week 6, Week 12 and Week 24.

ELIGIBILITY:
Inclusion Criteria:

1. Male or non-pregnant, non lactating females 18 years of age or older.
2. Signed informed consent form, which meets all criteria of current FDA regulations.
3. If female and of child bearing potential, have a negative urine pregnancy test at the baseline and randomization visits and prepared to abstain from sexual intercourse or use a reliable method of contraception during the study (e.g., condom with spermicide, inter-uterine device, oral, injected, transdermal or implanted hormonal contraceptives).
4. Clinical diagnosis of onychomycosis of at least one great toenail
5. Clinical signs and symptoms of onychomycosis of the most severely affected great toenail of at least moderate severity as defined by at least 25% but no more than 75% of the most infected toenail and a combined severity score of at least 4 using the Nail Infection Rating Scale (see Appendix A).
6. At least 2mm of clear nail on the most affected toe between the proximal nail fold and the deepest extend of the onychomycosis.
7. Positive potassium hydroxide (KOH) stain for confirmation of fungal nail infection
8. Positive mycological culture for known fungal dermatophyte consistent with onychomycosis infection of at least one of the great toenails.

Exclusion Criteria:

1. Females who are pregnant, lactating or likely to become pregnant during the study.
2. Negative KOH stain
3. Negative mycological culture for fungal dermatophytes consistent with onychomycosis infection.
4. Combined score of less than 4 on the Nail Infection Rating Scale for the most severely affected great toenail.
5. Patient has superficial onychomycosis or significant dystrophy of the target toenail that in the Investigators opinion would impair the evaluation of onychomycosis.
6. Patient has total dystrophic or proximal subungual onychomycosis of the target toenail.
7. Presence of mycotic spikes or patient has exclusively lateral groove involvement of the target toenail.
8. Less than 25% or more than 75% of the most severely infected great toenail affected.
9. Target toenail thickness is greater than 3mm.
10. No new nail growth in the target nail over the previous 6 months.
11. Onychomycosis not caused by a dermatophyte (e.g. mold infection, Candida spp or bacterial infection).
12. Previous treatment for onychomycosis of the toenail within the last 12 months that was unresponsive to treatment.
13. Previous treatment within the previous 2 months with any systemic antifungal therapy or within the previous 2 weeks with any topical antifungal therapy.
14. Significant history or current evidence of chronic infectious disease, system disorder, organ disorder or other medical condition that in the Investigator's opinion would place the study patient at undue risk by participation or could jeopardize the integrity of the study evaluations.
15. Immunocompromised either because of concomitant disease (e.g. HIV), or ongoing treatment (e.g. chemotherapy).
16. Current or history of psoriasis within the previous 12 months.
17. Evidence of ventricular dysfunction such as congestive heart failure (CHF) or a history of CHF.
18. History of diabetes.
19. Previous hypersensitivity to imidazole or azole compounds.
20. Liver Function Test results at screening more than twice the upper limit of normal range or other hematology or clinical chemistry test results that would contraindicate dosing with itraconazole.
21. Use within the previous 3 months or anticipated use during the study of any drugs that are known to affect the bioavailability of oral itraconazole or are otherwise contraindicated to be taken with itraconazole as detailed in the product labeling for SPORANOX® (Appendix B).
22. Receipt of any drug as part of a research study within 30 days prior to dosing.
23. Previous dosing in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 175 (Actual)
Dates: Start 2008-11; Primary Completion 2010-07 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Roger Aston, Study Chair — Halcygen Pharmaceuticals Limited
Locations (8):
- United States (8):
  - Synergyst Research, Altamonte Springs, Florida
  - FXM Research Corp, Miami, Florida
  - Northwest Clinical Trials, Boise, Idaho
  - PMG Research, Salisbury, North Carolina
  - Oregon Medical Research Center, P.C, Portland, Oregon
  - Coastal Carolina Research, Mt. Pleasant, South Carolina
  - JS Studies, College Station, Texas
  - Endeavor Clinical Trials, San Antonio, Texas

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo | Test | Reference
Started | 24 | 76 | 75
Completed | 19 | 60 | 61
Not Completed | 5 | 16 | 14

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Test | Reference | Total
Number analyzed (Participants) | 24 | 76 | 75 | 175
Age, Continuous [Mean (Full Range); unit: years of age] | 50.29 [21 to 73] | 47.41 [23 to 73] | 48.64 [21 to 78] | 48.78 [21 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 25 | 20 | 49
  Male | 20 | 51 | 55 | 126
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 0 | 1
  Black or African American | 2 | 1 | 6 | 9
  White | 21 | 74 | 69 | 164
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 24 | 76 | 75 | 175
Percentage of toe infected [Mean (Standard Deviation); unit: percentage] | 61.42 (15.99) | 55.08 (15.70) | 58.32 (14.99) | 58.27 (15.56)
Infecting organism - T.rubrum [Number; unit: participants] | 24 | 72 | 69 | 165
Presence of infecting organism - T.mentagrophytes [Number; unit: participants] | 0 | 3 | 6 | 9

OUTCOME MEASURES:

1. Primary Outcome: Non-inferiority Will be Determined by Evaluating the Difference Between the Proportion of Patients in the Test and Reference Treatment Groups Who Are Considered a "Therapeutic Cure" at the End of Study Visit (Week 24)
Description: If the lower bound 95% confidence interval of the difference between the proportion of patients in the Test group compared to the Reference group considered a Therapeutic Cure at Visit 7 was greater than 20 then non-inferiority was considered to have been demonstrated
Time Frame: Week 24
Population: The Efficacy evaluation was performed on the intent to treat population, which included all patients that met all the following criteria; positive baseline mycological culture, dosed with the study drug at least once and had at least one post-baseline evaluation
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Test | Reference
Number analyzed (Participants) | 24 | 76 | 74
Participants | 0 | 8 | 3
Statistical Analysis 1: Comparison: Test vs Reference; Test type: Non-Inferiority — To demonstrate non-inferiority an upper bound 95% confidence interval approach comparing the difference between the cure rate in the Test and the Reference groups was used. If the lower bound 95% confidence interval of the difference between the proportion of patients in the Test group compared to the Reference group considered a Therapeutic Cure, Clinical Cure and Mycological Cure as appropriate, at Week 24 was greater than -20 then non-inferiority was considered to have been demonstrated; -20 = 6.47, 95% CI 1-sided [lower limit -1.77]
Statistical Analysis 2: Comparison: Placebo vs Test; The ITT was used for all superiority testing. For the three primary endpoints and all four secondary endpoints, if the difference between the proportion of patients considered a cure was statistically greater (p<0.05) than the proportion of patients considered a cure in the Placebo group, then superiority was considered to have been demonstrated. A one-sided continuity corrected Z-test was used for superiority testing; Test type: Superiority; p < 0.05, one-sided continuity corrected Z-test

2. Primary Outcome: Non-inferiority Will be Determined by Evaluating the Difference Between the Proportion of Patients in the Test and Reference Treatment Groups Who Are Considered a "Clinical Cure" at the End of Study Visit (Week 24)
Description: If the lower bound 95% confidence interval of the difference between the proportion of patients in the Test group compared to the Reference group considered a Clinical Cure at Visit 7 was greater than 20 then non-inferiority was considered to have been demonstrated
Time Frame: Week 24
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Test | Reference
Number analyzed (Participants) | 24 | 76 | 74
Participants | 0 | 12 | 4
Statistical Analysis 1: Comparison: Test vs Reference; To demonstrate non-inferiority an upper bound 95% confidence interval approach comparing the difference between the cure rate in the Test and the Reference groups was used. If the lower bound 95% confidence interval of the difference between the proportion of patients in the Test group compared to the Reference group considered a Therapeutic Cure, Clinical Cure and Mycological Cure as appropriate, at Week 24 was greater than -20 then non-inferiority was considered to have been demonstrated; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; -20 = 10.38, 95% CI 1-sided [lower limit 0.92]
Statistical Analysis 2: Comparison: Placebo vs Test; [analysis description as in outcome 1, analysis 2]; Test type: Superiority; p < 0.05, one-sided continuity corrected Z-test

3. Primary Outcome: Non-inferiority Will be Determined by Evaluating the Difference Between the Proportion of Patients in the Test and Reference Treatment Groups Who Are Considered a "Mycological Cure" at the End of Study Visit (Week 24)
Description: If the lower bound 95% confidence interval of the difference between the proportion of patients in the Test group compared to the Reference group considered a Mycological Cure at Visit 7 was greater than 20 then non-inferiority was considered to have been demonstrated
Time Frame: Week 24
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Test | Reference
Number analyzed (Participants) | 24 | 76 | 74
Participants | 1 | 25 | 22
Statistical Analysis 1: Comparison: Test vs Reference; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; -20 = 3.17, 95% CI 1-sided [lower limit -10.62]
Statistical Analysis 2: Comparison: Placebo vs Test; [analysis description as in outcome 1, analysis 2]; Test type: Superiority; p < 0.05, one-sided continuity corrected Z-test

4. Secondary Outcome: The Proportion of Patients in Each Treatment Group Who Are Considered a "Therapeutic Cure" at the End of Treatment Visit (Week 12) 12).
Description: If the lower bound 95% confidence interval of the difference between the proportion of patients in the test group compared to the reference group considered a cure at the visit being analyzed was greater than -20 then non-inferiority was considered to have been demonstrated
Time Frame: Week 12
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Test | Reference
Number analyzed (Participants) | 24 | 76 | 74
Participants | 0 | 0 | 0

5. Secondary Outcome: Non-inferiority Will be Determined by Evaluating the Difference Between the Proportion of Patients in the Test and Reference Treatment Groups Who Are Considered a "Clinical Cure" at the End of Study Visit (Week 12)
Description: as for outcome 4
Time Frame: week 12
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Test | Reference
Number analyzed (Participants) | 24 | 76 | 74
Participants | 0 | 1 | 0

6. Secondary Outcome: Non-inferiority Will be Determined by Evaluating the Difference Between the Proportion of Patients in the Test and Reference Treatment Groups Who Are Considered a "Mycological Cure" at the End of Study Visit (Week 12)
Description: as for outcome 4
Time Frame: week 12
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Test | Reference
Number analyzed (Participants) | 24 | 76 | 74
Participants | 3 | 16 | 16
Statistical Analysis 1: Comparison: Test vs Reference; If the lower bound 95% confidence interval of the difference between the proportion of patients in the Test group compared to the Reference group considered a Therapeutic Cure, Clinical Cure or Mycological Cure as appropriate at Visit 7 was greater than -20 then non-inferiority was considered to have been demonstrated; Test type: Non-Inferiority — If the lower bound 95% confidence interval of the difference between the proportion of patients in the Test group compared to the Reference group considered a Therapeutic Cure, Clinical Cure or Mycological Cure as appropriate at Visit 7 was greater than -20 then non-inferiority was considered to have been demonstrated; -20 = -0.57, 95% CI 1-sided [lower limit -12.91]

7. Other Pre Specified Outcome: Superiority of Test Treatment Over Placebo for Mycological Cure
Description: All primary and secondary endpoints were tested for superiority against Placebo. The intent to treat (ITT) was used for all superiority testing. For the three primary endpoints and all four dichotomous secondary endpoints, if the difference between the proportion of patients considered a cure in the Test or Reference group was statistically greater (p < 0.05) than the proportion of patients considered a cure in the Placebo group, then superiority of that treatment over placebo was considered to have been demonstrated. A one-sided continuity corrected Z-test was used for superiority testing.
Time Frame: week 6
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Test | Reference
Number analyzed (Participants) | 24 | 76 | 74
Participants | 0 | 11 | 5
Statistical Analysis 1: Comparison: Placebo vs Test; For the three primary endpoints and all four dichotomous secondary endpoints, if the difference between the proportion of patients considered a cure in the Test or Reference group was statistically greater (p < 0.05) than the proportion of patients considered a cure in the Placebo group, then superiority of that treatment over placebo was considered to have been demonstrated. A one-sided continuity corrected Z-test was used for superiority testing; Test type: Superiority; p < 0.05, A one-sided continuity corrected Z-test — It the difference between the proportion of patients considered a cure was statistically greater (p<0.05) than the proportion of patients considered a cure in the Placebo group, then superiority was considered to have been demonstrated; Mean Difference (Final Values) = 0.0018
Statistical Analysis 2: Comparison: Placebo vs Reference; [analysis description as in outcome 7, analysis 1]; Test type: Superiority; p < 0.05, A one-sided continuity corrected Z-test; Median Difference (Final Values) = 0.0853

ADVERSE EVENTS:
Time Frame: The safety profile of each treatment group was evaluated by comparing adverse events, monitoring vital signs, EKG parameters, audiology testing, and changes in clinical laboratory results obtained throughout the study, which included the 12 week treatment period and the End of Study Visit at Week 24.
Arm/Group | Placebo | Test | Reference
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/76 | 0/75
Serious Adverse Events (participants affected / at risk) | 0/24 | 2/76 | 1/75
Other Adverse Events (participants affected / at risk) | 13/24 | 42/76 | 35/75
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=24) | Test (N=76) | Reference (N=75)
Pulmonary Embolism (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) — Possibly related
Lumbar Spinal Stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) — Unrelated
Intervertebral disc protusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) — Unrelated
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=24) | Test (N=76) | Reference (N=75)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Acoustic Stimulation Tests Abnormal (Ear and labyrinth disorders) | 0 (0) | 2 (2) | 3 (3)
Alanine Aminotransferase Increased (Investigations) | 0 (0) | 3 (3) | 2 (2)
Arthropod Bite (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Aspartate Aminotransferase Increased (Investigations) | 0 (0) | 3 (3) | 1 (1)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 3 (3)
Depressed Mood (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Dermatitis Contact (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Erectile Dysfunction (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Gastroesophageal Reflux Disease (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 2 (2) | 7 (7) | 8 (8)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 1 (1) | 2 (2)
Insomnia (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0)
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2)
Nasopharyngitis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 7 (7) | 5 (5)
Nausea (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Ooropharyngeal Pain (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 4 (4)
Rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 0 (0)
Sinus Headache (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0)
Sinusitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 0 (0)
Tension Headache (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 2 (2)
Upper Respiratory Tract Congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Upper Respiratory Tract Infection (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 3 (3)
Vertigo (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Subjects were followed for 12 weeks after the 12 week treatment period, typically subjects would be followed for at least 24 weeks post-treatment to allow sufficient time for the nail to grow out and therefore maximizing rates of clinical cure

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less